CLINICAL TRIAL: NCT01604239
Title: A 24 Weeks, Multi-centers, Single Arm Phase IV Study to Evaluate the Safety of 'Shinbaro Capsule' Compared With Historical Data of 'Celebrex Capsule' in Patients With Osteoarthritis
Brief Title: To Evaluate the Safety of 'Shinbaro Capsule'in Patients With Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCSB_P4
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Shinbaro; Herbal drug
MeSH Terms: conditions — Osteoarthritis | interventions — shinbaro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Shinbaro (Experimental)
  Interventions: Drug: Shinbaro Capsule

INTERVENTIONS:
Drug: Shinbaro Capsule — 600mg twice a day (b.i.d) oral herbal medicine

SUMMARY:
This study investigates if Shinbaro capsule has a lower incident of gastrointestinal events than celecoxib in subjects with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 19 years old
* Kellgren stage I ~ III by ACR criteria
* Stable osteoarthritis during 3 months
* Be able to perform WOMAC and KKS
* Written consent form voluntarily

Exclusion Criteria:

* Disease of orthopaedic surgical that could affect to evaluate the efficacy
* Medication of continuous corticosteroid by oral or articular cavity within 12 weeks
* Medication of constantly (more than 1 week) antipsychotic drug or narcotic analgesics within four weeks
* Medical history of hypersensitivity reaction against Herbal drug
* Genetic factors as galactose intolerance, lapplactase deficiency or glucose-galactose malabsorption, etc.
* Occurrence of OA caused by the injury
* Diagnosed with psychical disorder, and taking medication
* Diagnosed with active peptic ulcers, gastrointestinal bleeding, inflammatory bowel disease, severe liver dysfunction, severe renal dysfunction, congestive heart failure, clinically significant ischemic heart disease, peripheral arterial disease, or cerebrovascular diseases
* Diagnosed with esophagus and gastrointestinal ulceration within 1 year, or treated it
* Abnormal bleeding (abnormal of platelet or blood coagulation factor, etc.)
* Positive in fecal occult blood test
* Gastrointestinal tract surgery except appendectomy
* Serum creatinine, ALT, AST, total bilirubin over UNL x 1.5 at screening test
* Participation in another clinical trials within 4 weeks
* Not consent about using effectual contraception method during trial
* Pregnant or lactating woman
* Medical history of malignant tumor within 5 years
* Investigator's judgment

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 761 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with gastrointestinal adverse events | Baseline through 24 weeks

SECONDARY OUTCOMES:
percentage of subjects with perforation, ulcer, bleeding | baseline throgh week 24
percentage of subjects who withdrew due to GI AEs | baseline through week 24
Frequency of AEs | baseline throgh week 24
WOMAC change from baseline | 24 weeks
KKS (Korean Knee Score) change from baseline | 24 weeks
100mm pain VAS on walking | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: BG Lee, Study Chair — GC Biopharma Corp
Locations (18):
- South Korea (18):
  - Kyungpook national university hospital, Daegu, Kyungpook
  - BundangCha Hospital, Bundang
  - Inje University Busan Paik Hospital, Busan
  - Chungbuk National University Hospital, Cheongju-si
  - Keimyung University Dongsan Medical Center, Daegu
  - Yeungnam University Hospital, Deagu
  - Chonnam National University Hwasun Hospital, Hwasun
  - Dongguk University Medical Center, Ilsan
  - Inha University Hospital, Inchun
  - Chonbul National University Hospital, Jeonju
  - Samsung Medical Center, Seoul
  - Asan medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Inje University Seoul Paik Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Ha CW, Park YB, Kyung HS, Han CS, Bae KC, Lim HC, Park SE, Lee MC, Won YY, Lee DC, Cho SD, Kim CW, Kim JG, Kang JS, Lee JH, Choi ES, Seon JK, Lee WS, Bin SI. Gastrointestinal safety and efficacy of long-term GCSB-5 use in patients with osteoarthritis: A 24-week, multicenter study. J Ethnopharmacol. 2016 Aug 2;189:310-8. doi: 10.1016/j.jep.2016.05.031. Epub 2016 May 16. PMID 27196293